CLINICAL TRIAL: NCT01102556
Title: PREDICT: Pancreatic Disease Cohort. A Registry and Biospecimen Bank To Better Understand Pancreatic Disease.
Brief Title: PANCREATIC DISEASE COHORT A Registry and Biospecimen Bank to Better Understand Pancreatic Disease
Status: Recruiting | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Other Study IDs: AAAA6154
Record Dates: First submitted 2010-04-12; First posted 2010-04-13 (Estimated); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer; Pre-Neoplastic Lesions; Pancreatic Cancer Surgery; High-Risk for Pancreatic Cancer; Tissue and Blood Bank for Pancreatic Cancer; Pancreatic Cancer Questionnaire
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — * Peripheral Blood Specimens: Three tubes of blood will be collected from each study participant.
  * Archived Fixed Tissue Samples: Tissue blocks from surgery performed at CUMC or elsewhere, will be requested after obtaining consent for study participation.
  * Fresh Tissue Collection: At the time of surgery for any tumor resection, tumor tissue and adjacent normal tissue will be requested from the Pathology Department. At the time of endoscopy, aspirated fluid or biopsied tissue will be requested. No additional tissue will be resected beyond that required for surgical or endoscopic management. In no circumstance will tissue be obtained solely for the purpose of the study.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Surgery Patients/High-risk Patients: Patients who have undergone surgery for pancreatic cancer or pre-neoplastic lesions of the pancreas will be accrued to the study. In addition, patients who are determined to be at high-risk for pancreatic cancer (with a significant family history) will also be recruited for study enrollment.

SUMMARY:
The specific aims of this project are to create a registry, as well as a biospecimen bank for individuals with pancreatic disease (e.g. pancreatic adenocarcinoma, pancreatitis, intraductal papillary mucinous neoplasm (IPMN) mucinous cystic neoplasm (MCN), and pancreatic intraepithelial neoplasia (PanIN) or have been determined to be at high-risk for pancreatic cancer. Biospecimen can be defined as blood, urine, tissue, stool, or saliva samples. Therefore, no hypothesis is to be tested. The personal data derived from the registry, correlated with biological information derived from the biospecimens will allow for future investigative studies of pancreatic cancer etiology and tumor biology. The long-term goals of the study are to advance the knowledge of the etiology and epidemiology of pancreatic cancer. It is anticipated that the knowledge derived will ultimately lead to improvements in the diagnosis, prevention, detection,and treatment of pancreatic cancer.

DETAILED DESCRIPTION:
Pancreatic cancer is the fourth leading cause of cancer death in both men and women in the United States. According to the American Cancer Society facts and figures, approximately 43,920 people in the United Sates will be diagnosed with pancreatic cancer in 2012, and it is expected that 37,390 will die from the disease. The dismal prognosis of the disease is clearly depicted by the fact that its incidence approximates its mortality. Pancreatic cancer has a 95% case fatality rate. The etiology of pancreatic cancer remains elusive and our knowledge of its precursors and natural history is preliminary and incomplete. The uniform fatality of the disease merits priority attention in the search for its cause.

Due to the rapid progression of the disease, early detection and prevention provides the best hope for reducing morbidity and mortality. However, the few screening tests available for early detection and/or prevention of neoplastic lesions are poorly studied and prohibitively impractical in the general population. Further, few pancreatic cancer risk factors are well established or widely accepted. Advanced age, family history, cigarette smoking, diabetes, and some dietary risk factors are established or suspected risk factors.

Due to the high volume of individuals seen at the pancreas center, we plan on enrolling 500+ individuals per year who have either been diagnosed with pancreatic disease or are at high risk for developing pancreatic cancer. All participants enrolled during a clinic/non clinic visit at Columbia University Medical Center (CUMC) will undergo a baseline visit and up to 3 subsequent visits. Additionally, based on the different conditions of pancreatic disease that we are enrolling, not all subjects will participate in all aspects of the program. For example, only individuals with cancer or pre-neoplastic lesions will have tissue collected and banked.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have been diagnosed with pancreatic cancer or suspicion of pancreatic cancer, a pre-neoplastic lesion in the pancreas who are 18 years or older
* Individuals identified to be high risk for developing pancreatic cancer who are 18 years or older based on the following criteria:
* The modified clinical Bethesda criteria for hereditary nonpolyposis colorectal cancer (HNPCC), which are as follows: individuals with 2 HNPCC-associated cancers (colon, endometrial, small bowel, hepatobiliary, pancreatic, genitourinary, or gastric), including synchronous or metachronous lesions; individuals with colon cancer and a first degree relative with an HNPCC-associated tumor and/or colonic adenoma (1 cancer diagnosed at age <45 years and the adenoma diagnosed at age <40 years); individuals with colon or endometrial cancer diagnosed at <50 years; individuals with right-sided colon cancer having an undifferentiated pattern (solid/cribiform) or signet cell histopathology diagnosed at <45 years; or individuals with adenomas diagnosed at <40 years.
* Those with a personal or family history of other pancreatic cancer associated syndromes including: Peutz-Jeghers syndrome, familial pancreatic cancer syndrome, familial breast cancer syndrome associated with BReast CAncer genes 1 or 2 (BRCA-2 or BRCA-1), hereditary pancreatitis, familial atypical multiple mole melanoma, and others.
* Patients in a family with a genetically determined cancer predisposition syndrome.
* Patients with a personal history of a gastrointestinal malignancy at age <45 years.
* Individuals at high-risk based on personal or family history, but not related to a known pancreatic cancer syndrome include the following: those with a personal history of pancreatic cancer, or a pre-neoplastic pancreatic lesion; those with a family history of two or more individuals with cancer, at least one of which is reported to be a gastrointestinal malignancy; a history of early onset (<50 years) gastrointestinal cancer in the individual or a family member; a history of multiple primary cancers, at least one of which is a gastrointestinal primary, or a family member of an individual meeting this criterion.

Exclusion Criteria:

* Inability to obtain informed consent for study enrollment.
* Under the age of 18 years old.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals who have been diagnosed with pancreatic cancer or suspicion of pancreatic cancer, a pre-neoplastic lesion in the pancreas, or who have been identified to be at high-risk for developing pancreatic cancer.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2004-07 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Creation of a registry and blood/tissue bank | 1 year
  The primary aims of this project are to create a registry, and blood and tissue bank for individuals at risk for pancreatic cancer.

SECONDARY OUTCOMES:
Improvement in the diagnosis, prevention, detection, and treatment of pancreatic cancer. | 10 years
  The long-term goals of the study are to advance the knowledge of the etiology and epidemiology of pancreatic cancer. The epidemiological data will be correlated with the biological information and will allow for future investigative studies of pancreatic cancer etiology and tumor biology. It is anticipated and hypothesized that the knowledge derived will lead to improvements in the diagnosis, prevention, detection, and treatment of pancreatic cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Beth Schrope, MD, PhD, FACS, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No